CLINICAL TRIAL: NCT00125021
Title: A Phase II Study of OSI-774 (Tarceva) in Combination With Capecitabine in Previously Treated Patients With Metastatic Pancreatic Cancer
Brief Title: Tarceva and Capecitabine for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Roche Global Development (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Matthew Kulke, MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-070
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Pancreatic Cancer; Neoplasm Metastasis
Keywords: Second Line Therapy; Gemcitabine Refractory; Pancreatic Cancer; Capecitabine; Tarceva; OSI-774; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Capecitabine — Given twice a day for 14 days followed by 7 days of no capecitabine (1 cycle is 21 days).
Drug: OSI-774 — Given once daily
  Other Names: Tarceva

SUMMARY:
This phase II trial is designed to investigate the effectiveness of Tarceva (OSI-774) combined with capecitabine in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Patients will be treated once daily with Tarceva, twice daily with capecitabine for 14 consecutive days, followed by 7 days off of capecitabine (a cycle is 21 days). At week 1 of each cycle a physical exam and blood work will be performed. Reassessment of tumor size will be conducted at 6 weeks (2 cycles), 12 weeks (4 cycles) and then every 9 weeks thereafter. Patients will remain on treatment until one of the following occur: disease progression, illness that prevents further treatment or unacceptable adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic carcinoma (excluding pancreatic endocrine tumors)
* Only patients with measurable disease
* ECOG performance status < or equal to 1
* Life expectancy >12 weeks
* Signed informed consent
* Failed or intolerance to first-line therapy for metastatic disease with a gemcitabine-containing regimen. Patients may have received adjuvant therapy in addition to one prior regimen for metastatic disease.
* >4 weeks must have elapsed from the completion of previous chemotherapy and patients must have recovered from any related toxicities
* >4 weeks must have elapsed from the participation in any investigational drug study
* Laboratory values:

  * ANC > 1500/mm3;
  * Hemoglobin > 9.0 gm/dl;
  * Platelets > 100,000/mm3;
  * SGOT <2.5 X upper limit of normal; or <5 X upper limit of normal if evidence of liver metastases; Alkaline phosphatase < 2.5 X upper limit of normal; or < 5 X upper limit of normal if evidence of liver metastases; Total bilirubin < 1.5 X upper limit of normal; Creatinine clearance > 50 cc/min (by Cockroft - Gault or as determined from a 24-hour urine collection).

Exclusion Criteria:

* Prior therapy with capecitabine or epidermal growth factor receptor (EGFR) inhibitors
* More than one prior chemotherapy treatment regimen for metastatic disease
* Clinically apparent central nervous system (CNS) metastases or carcinomatous meningitis
* Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication or heart attack within the last 12 months).
* Major surgery within 4 weeks of the start of study treatment, without complete recovery.
* Evidence of CNS metastases (unless CNS metastases have been stable for > 3 months) or history of uncontrolled seizures, central nervous system disorders
* Uncontrolled serious medical or psychiatric illness
* Women must not be pregnant or lactating
* Concurrent radiation therapy
* Other active malignancy
* Inability to swallow tablets
* Patients lacking physical integrity of the upper gastrointestinal tract or who have malabsorption syndrome
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-10; Primary Completion 2004-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To assess the response rate associated with capecitabine and OSI-774 in patients with advanced pancreatic cancer

SECONDARY OUTCOMES:
To assess the side effects of capecitabine and OSI-774 in patients with advanced pancreatic cancer | 2 years
to estimate the time to progression and overall survival of patients with advanced pancreatic cancer treated with capecitabine and OSI-774

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kulke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts